CLINICAL TRIAL: NCT04306484
Title: 18F-DOPA-PET in Non-tumoral and Tumoral Brain Lesions
Acronym: FDOPA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2020/DR-01
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2020-03

CONDITIONS: Brain Tumor
Keywords: tumor; tumoral; non-tumoral; pseudotumoral; 3,4-dihydroxy-6-[18F]-fluoro-L-phenylalanine; FDOPA; positron emission tomography; PET
MeSH Terms: conditions — Brain Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with tumoral brain lesion: The 48 tumor patients included 8 low grade (grade II glioma, n=7; grade II ependymoma, n=1), and 40 high grade (grade III glioma, n=12; grade IV glioma, n=25, primary cerebral lymphoma, n=1; medulloblastoma, n=1, and metastatic cerebral breast cancer, n=1) tumors. Histology was available for all tumor patients.
  Interventions: Diagnostic Test: FDOPA-TEP
- patients with non-tumoral brain lesion: The non-tumor group included patients with an inflammatory lesion (n=11), lobar primary intracerebral haemorrhage (n=3), cortical dysplasia (n=3), infectious lesion (n=2, both toxoplasmosis), cerebral cavernomatous malformation (n=1), seronegative autoimmune limbic encephalitis (n=1), deep venous sinus thrombosis-related oedema (n=1), brain infarction (n=1), chronic posttraumatic brain lesion (n=1), radionecrosis after radiation therapy for arteriovenous malformation (n=1), and mixed inflammatory/infectious lesion (n=1, multiple sclerosis lesion complicated by biopsy-related infection).
  Interventions: Diagnostic Test: FDOPA-TEP

INTERVENTIONS:
Diagnostic Test: FDOPA-TEP — FDOPA-TEP performed as part of the normal management of a suspected brain tumour

SUMMARY:
Background: 3,4-dihydroxy-6-[18F]-fluoro-L-phenylalanine (FDOPA) positron emission tomography (PET) can identify well low and high grade brain tumors. However, increased FDOPA uptake has been reported in non-tumoral brain lesions. The aim was to analyse FDOPA-PET in patients with non-tumoral brain lesions and to compare them with patients with (low and high grade) brain tumors.

Methods: retrospective analyse. Patients consecutively recruited with suspected primary brain tumor (based on clinical and MRI findings) referred for FDOPA-PET at Nimes university Hospital between June 2015 and June 2019. FDOPA-PET parameters (maximum and mean lesion standardized uptake values [SUV] and ratios comparing lesion with different background uptake SUV) and thresholds were analysed in search for those offering optimal discrimination between non-tumoral and tumoral lesions.

ELIGIBILITY:
Inclusion Criteria:

* presence of defined tumor (histology was required) or non-tumor (diagnosed by histological or other analyses) diagnosis,
* clinical and MRI follow-up of >24 months,
* FDOPA-PET scan <2 months before surgery or stereotactic biopsy (when performed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected primary brain tumor (based on clinical and MRI findings) referred for FDOPA-PET in our centre between June 2015 and June 2019
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
FDOPA-TEP | Day 1
  analyse of FDOPA-PET parameters (maximum and mean lesion standardized uptake values [SUV] and ratios comparing lesion with different background uptake SUV)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Renard D, Collombier L, Laurent-Chabalier S, Mura T, Le Floch A, Fertit HE, Thouvenot E, Guillamo JS. 18F-FDOPA-PET in pseudotumoral brain lesions. J Neurol. 2021 Apr;268(4):1266-1275. doi: 10.1007/s00415-020-10269-9. Epub 2020 Oct 21. PMID 33084938